CLINICAL TRIAL: NCT01139320
Title: Pharmacogenetics of Mylotarg
Brief Title: Biomarkers in DNA Samples From Younger Patients With Newly Diagnosed Acute Myeloid Leukemia Receiving Gemtuzumab Ozogamicin
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B3; COG-AAML10B3 (Other: Children's Oncology Group); CDR0000671448 (Other: Clinical Trials.gov); NCI-2011-02220 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-05; First posted 2010-06-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of DNA from patients receiving gemtuzumab ozogamicin may help doctors learn more about the effects of gemtuzumab ozogamicin on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers in DNA samples from younger patients with newly diagnosed with acute myeloid leukemia receiving gemtuzumab ozogamicin.

DETAILED DESCRIPTION:
OBJECTIVES:

* To analyze candidate-coding polymorphisms in CD33 of DNA samples from children with newly diagnosed acute myeloid leukemia treated with gemtuzumab ozogamicin on COG-AAML03P1.
* To determine the association between these polymorphisms and clinical response of patients treated with this regimen.

OUTLINE: Archived DNA samples are analyzed for candidate polymorphisms in CD33 by PCR-based sequencing.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia
* Treated with gemtuzumab ozogamicin on COG-AAML03P1
* Genomic DNA samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed acute myeloid leukemia treated with gemtuzumab ozogamicin on COG-AAML03P1.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Association between coding polymorphisms in CD33 with clinical response to gemtuzumab ozogamicin

CONTACTS AND LOCATIONS:
Overall Officials: Jatinder Lamba, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota